CLINICAL TRIAL: NCT07278349
Title: Randomized, Single Dose, Two-Way Crossover, Open Label Bioequivalence Study to Compare Vonoprazan 20 mg Film Coated Tablets Versus Voquezna® 20 mg (Vonoprazan) Tablets an Oral Administration to Healthy Adults Under Fasting Conditions
Brief Title: Bioequivalence Study to Compare Vonoprazan 20 mg Film Coated Tablets Versus Voquezna® 20 mg (Vonoprazan) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VON-T003
Record Dates: First submitted 2025-12-09; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Erosive Gastritis; Erosive Esophagitis(EE); HELICOBACTER PYLORI INFECTIONS
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VONOPRAZAN FILM COATED TABLETS (Experimental): VONOPRAZAN FILM COATED TABLETS (20 mg Vonoprazan)
  Interventions: Drug: Vonoprazan Tablets; Drug: VOQUEZNA® Tablets
- VOQUEZNA® (VONOPRAZAN) TABLETS (Active Comparator): VOQUEZNA® (VONOPRAZAN) TABLETS (20 mg Vonoprazan)
  Interventions: Drug: Vonoprazan Tablets; Drug: VOQUEZNA® Tablets

INTERVENTIONS:
Drug: Vonoprazan Tablets — 1 tablet of 20 mg Vonoprazan
Drug: VOQUEZNA® Tablets — 1 tablet of 20 mg Vonoprazan

SUMMARY:
Randomized, Single Dose, Two-Way Crossover, Open Label bioequivalence study to compare Vonoprazan 20 mg Film Coated Tablets versus Voquezna® 20 mg (Vonoprazan) Tablets an oral administration to healthy adults under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant, age 18 to 50 years, inclusive.
* Body Mass Index (BMI) range5 is within 18.5 - 30 Kg/m2.
* Participant does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.
* Standard ECG assessment is normal and no QTc Prolongation (QTc ≤ 450 ms in male and QTc ≤ 460 ms in females).
* Medical history and physical examination within medically acceptable criteria.
* Participant is capable of consent.

Exclusion Criteria:

* Demographics data with significant deviations from the normal ranges.
* Presence of any clinically significant results from laboratory reference ranges, however, ALP and creatinine will be accepted if below reference range after being evaluated by the physician as clinically not significant. RBC count, PCV, MCV, MCH and MCHC with deviation of more than 5% of the reference limits for all laboratory tests that are performed not longer than two weeks before the initiation of the clinical study.
* History of drug or alcohol abuse.
* Participant is a heavy smoker (more than 10 cigarettes per day).
* Participant does not agree to not taking any prescription or non-prescription drugs within at least two weeks before first study drug administration and until donating the last sample of the study.
* Participant does not agree to not taking any vitamins taken for nutritional purposes within at least two days before first study drug administration and until donating the last sample of the study.
* Participant is on a special diet (for example participant is vegetarian).
* Participant consumes large quantities of alcohol or beverages containing methyl-xanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc.).
* Participant does not agree to not consuming any beverages or food containing alcohol at least 2 weeks prior to first study drug administration until donating the last sample of the study.
* Participant does not agree to not consuming any beverages or food containing methyl-xanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc.) at least 24 hours prior to the study drug administration of either study periods until the end of confinement.
* Participant does not agree to not consuming any beverages or food containing grapefruit at least 2 weeks prior to first study drug administration until donating the last sample of the study.
* Participant has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 80 days before first study drug administration.
* Participant intends to be hospitalized within 3 months after first study drug administration.
* Participants who donated blood or its derivatives in the past 3 months or who through completion of this study, would have donated more than 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.
* Participant has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders.
* Participant does not agree to not be engaged in strenuous exercise at least one day prior to study drug administration until donating the last sample in each respective period.
* Participant having at screening examination a pulse outside the normal range of (60-100 beats per minute) or a body temperature outside the normal range of (35.0-37.2 °C) or a respiratory rate outside the normal range of (12-20 breaths per minute) or a sitting blood pressure less than 100/60 mm Hg or more than or equal to 140/90 mm Hg.
* Participant has history of difficulties in swallowing or any gastrointestinal disease which could affect the drug absorption.
* Positive blood screen for HIV, Hepatitis B surface antigen (HBsAg), or Hepatitis C.
* Participant has a difficulty fasting or consuming standard meals.
* The participant is a pregnant or lactating female.
* Participant does not agree to not consuming any medication or food which may affect CYP3A4/5, CYP2B6, CYP2C19, CYP2C9 and CYP2D6 enzymes at least two weeks prior to first study drug administration until donating the last sample of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-09-21 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximal Plasma Concentration) | 48.00 hours
  The point estimate and the 90% confidence intervals of the mean values for the Test/Reference ratio were within the bioequivalence acceptable boundaries of 80.00-125.00%
AUC0-t (Area Under the plasma concentration-time Curve from zero (0) hours to time (t) hours) | 48.00 hours
  The point estimate and the 90% confidence intervals of the mean values for the Test/Reference ratio were within the bioequivalence acceptable boundaries of 80.00-125.00%

SECONDARY OUTCOMES:
AUC0-∞ (Area Under the plasma concentration-time Curve from zero (0) hours to infinity (∞)) | 48.00 hours
  Descriptive statistics
Kel (Elimination Rate Constant ) | 48.00 hours
  Descriptive statistics
tmax (Time until maximum plasma concentration is reached ) | 48.00 hours
  Descriptive statistics
t½el (Plasma concentration half-life) | 48.00 hours
  Descriptive statistics

CONTACTS AND LOCATIONS:
Locations (1):
- IPRC International Pharmaceutical Research Center, Amman, Sport City Circle, Jordan

IPD SHARING:
Plan to Share IPD: No